CLINICAL TRIAL: NCT05843071
Title: An Interventional, Non-comparative, Single-center Post Marketing Clinical Follow-up (PMCF) Study to Evaluate Performance and Safety of "NASAL SPRAYS " Used to Relieve Nasal Congestion and Dryness
Brief Title: PMCF Study to Evaluate Performance and Safety of "NASAL SPRAYS " Used to Relieve Nasal Congestion and Dryness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C.O.C. Farmaceutici S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COC-R8-NS
Record Dates: First submitted 2023-04-13; First posted 2023-05-06 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2023-05

CONDITIONS: Nasal Congestion; Nasal Dryness
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nasal spray treatment arm (Experimental)
  Interventions: Device: Nasal sprays with sea salts

INTERVENTIONS:
Device: Nasal sprays with sea salts — Nasal sprays for nasal congestion and dryness

SUMMARY:
Acute viral upper respiratory tract infection, also known as common cold, is the most frequently observed infectious disease in human beings. Although common cold is a self-limiting disease, symptoms such as runny nose, nasal congestion, sneezing, cough, sore throat, are troublesome.

Dry nose is characterized by nasal mucosa dryness, itching, mild burning, crusting, and dehydrated mucus. Causes of dry nose sensation include climatic factors, dry room air, workplace conditions, allergic rhinitis, endonasal sinus surgery.

Dry nose symptoms occur concurrently and may be the first signs of a common cold infection and rhinitis sicca (also known atrophic rhinitis).

Saline nasal sprays are broadly used as first-line treatment to relieve nasal congestion or nasal dryness. Isotonic saline solutions preferentially aim at cleansing and moistening of the nasal mucosa and thus are suitable for treatment of dry nose symptoms. Hypertonic saline solutions are generally used for decongestion of the nasal mucosa.

For these reasons, an interventional, non-comparative, single-center Post Marketing Clinical Follow-up (PMCF) study was planned to evaluate the performance and safety of "NASAL SPRAYS" used to relieve nasal congestion and dryness.

The objectives of the PMCF study are confirmation of the performance, collection of additional safety data regarding expected adverse events and detection of potential unexpected adverse events associated with the use of "NASAL SPRAYS" according to the instruction for use (IFU).

Each pediatric subject whose parent(s)/legal guardian signed an Informed Consent Form (ICF), and each adult subject after signing the ICF, will enter the screening and baseline phase (the 2 visits will coincide) during which baseline procedures will be completed.

At baseline visit (V0), one of the "NASAL SPRAYS" will be administered to the enrolled subject.

The patient will perform 2 on-site visits: V0 and V2/EOS. To monitor the safety, 1 phone contact is planned (V1) to check for potential adverse events and concomitant medications intake.

The first administration and the intervals at which the treatment should be repeated, to be done as per Investigator judgment and according to the IFU, depend on various factors regarding the physiology of the patients (e.g. nasal congestion/ obstruction, sneezing), the age of the patient, and for pediatric subjects, their birth characteristics (e.g. age, prematurity, birthweight).

ELIGIBILITY:
Inclusion Criteria:

* Pediatric subjects whose ICF will be signed by parent(s) or legal guardian;
* Adults' ICF signed;
* M & F infants (6-23 months), children (2-11 years), or M & F Aged ≥ 18 years at the time of the signature of the ICF;
* Infants, children or adults presenting with nasal congestion and/or nasal dryness.
* Willingness not to use other nasal sprays during the entire study.

Exclusion Criteria:

* Suspected other - different - conditions involving the respiratory tract (e.g. asthma, pneumonia);
* Suspected or known hypersensitivity or allergy to Investigational Product (IP) components;
* Suspected alcohol or drug abuse;
* Other clinically significant and uncontrolled pathologies that may interfere with study results (e.g. cystic fibrosis);
* Participation in another investigational study;
* Parent(s)' and/or patient's inability to follow all study procedures, including attending all site visits, tests and examinations;
* Parent(s)' and/or patient's mental incapacity that precludes adequate understanding or cooperation.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-06-19 (Actual)

PRIMARY OUTCOMES:
Change in nasal symptoms:To evaluate the performance of the "NASAL SPRAYS" used to relieve nasal congestion and dryness, through Visual Analogue Scale (VAS) for assessment of nasal symptoms | From baseline (V0 = Day 0) to 10 days (EOS/V2 - Day 10 ± 1)
  Visual Analogue Scale:
  Minimum value = 0; Maximum value = 10; Higher scores mean a better outcome.

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of the "NASAL SPRAYS" through visual nasal examination and assessment of AEs including the relationship of the AE to the IP (e.g. local allergic reaction) | End of study visit (EOS/V2 - Day 10 ± 1)
Change in Quality of life: to evaluate the capability of the "NASAL SPRAYS" to improve the (QoL), through Visual Analogue Scale (VAS) for assessment of QoL | End of study visit (EOS/V2 - Day 10 ± 1)
  Visual Analogue Scale:
  Minimum value = 0; Maximum value = 10; Higher scores mean a better outcome.
To evaluate the parent(s), children or adults' satisfaction of the "NASAL SPRAYS" through a 5-points Likert scale | End of study visit (EOS/V2 = Day 10 ± 1)

CONTACTS AND LOCATIONS:
Locations (1):
- U.O.C otorinolaringoiatria, Policlinico Mater Domini, Catanzaro, CZ, Italy